CLINICAL TRIAL: NCT03029754
Title: Effect of Passive Leg Raise for Pediatric Peripheral IV Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio 16-331
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Intravenous Access

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive leg raise (Experimental): Participant's legs will be raised with a bolster prior to IV insertion.
  Interventions: Procedure: Passive leg raise
- No leg raise (No Intervention): Participants will lie flat prior to IV insertion.

INTERVENTIONS:
Procedure: Passive leg raise — A baseline vein diameter will be obtained using ultrasound by the sub-investigator. Then a nurse will raise the child's legs using a bolster while a second measurement of the child's vein diameter is recorded by the sub-investigator. The anesthesiologist will then place the IV and rate the degree of difficulty encountered.
  Arms: Passive leg raise

SUMMARY:
The investigators wish to determine whether passive leg raise allows for easier peripheral vascular access in the pediatric population. The investigators hypothesize that pediatric anesthesiologists will have higher rates of successful intravenous catheterization in children where a passive leg raise is employed.

ELIGIBILITY:
Inclusion Criteria:

* pediatric participants undergoing dental procedures under general anesthesia

Exclusion Criteria:

* Children who already have adequate IV access

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Mean change in peripheral vein diameter | at 5 minutes
  Change between vein diameter at baseline and following group allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Gamble, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No